CLINICAL TRIAL: NCT00086879
Title: Randomized Phase II of TARCEVA™ (Erlotinib) Versus Temozolomide Or BCNU in Patients With Recurrent Glioblastoma Multiforme
Brief Title: Erlotinib Compared With Temozolomide or Carmustine in Treating Patients With Recurrent Glioblastoma Multiforme
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-26034-16031; EORTC-26034-16031
Record Dates: First submitted 2004-07-08; First posted 2004-07-12 (Estimated); Last update posted 2017-07-27 (Actual); Status verified 2017-07

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult glioblastoma; recurrent adult brain tumor; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Glioblastoma; Brain Neoplasms; Gliosarcoma | interventions — Carmustine; Erlotinib Hydrochloride; Temozolomide

INTERVENTIONS:
Drug: carmustine
Drug: erlotinib hydrochloride
Drug: temozolomide

SUMMARY:
RATIONALE: Erlotinib may stop the growth of tumor cells by blocking the enzymes necessary for their growth. Drugs used in chemotherapy, such as temozolomide and carmustine, work in different ways to stop tumor cells from dividing so they stop growing or die. It is not yet known whether erlotinib is more effective than temozolomide or carmustine in treating recurrent glioblastoma multiforme.

PURPOSE: This randomized phase II trial is studying erlotinib to see how well it works compared to temozolomide or carmustine in treating patients with recurrent glioblastoma multiforme.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the therapeutic activity of erlotinib vs temozolomide or carmustine in patients with recurrent glioblastoma multiforme.
* Compare 6-month progression-free survival in patients treated with these drugs.

Secondary

* Compare the safety of these drugs in these patients.

OUTLINE: This is a randomized, open-label, multicenter study. Patients are stratified according to participating center. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral erlotinib* once daily on day 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

NOTE: *Patients treated with enzyme inducing anti-epileptic drugs (EIAEDs) receive a higher dose of erlotinib than patients not receiving any anti-epileptic drugs or EIAEDs.

* Arm II: Patients who have not received prior temozolomide are assigned to receive temozolomide. Patients who have received prior temozolomide are assigned to receive carmustine. Patients receive 1 of the following treatment regimens:

  * Patients receive oral temozolomide* once daily on days 1-5. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  * Patients receive carmustine IV once daily on days 1-3. Treatment repeats every 56 days for up to 5 courses in the absence of disease progression or unacceptable toxicity.

NOTE: *Chemotherapy-naïve patients receive a higher dose of temozolomide than patients who have received prior adjuvant chemotherapy.

Patients are followed every 8 weeks until disease progression and then every 3 months thereafter.

PROJECTED ACCRUAL: A total of 100-110 patients (50-55 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed glioblastoma multiforme

  * Some oligodendroglial elements allowed provided they make up < 25% of the tumor
* Recurrent disease documented by MRI after prior radiotherapy
* At least 1 bidimensionally measurable target lesion ≥ 2 cm by MRI
* Undergone prior surgery for recurrent primary brain tumor more than 3 months before study entry

  * Must have a clearly limited target lesion ≥ 2 cm OR evidence of progressive and measurable target lesion OR a second measurable target lesion outside the surgical area

PATIENT CHARACTERISTICS:

Age

* Over 18

Performance status

* Karnofsky 70-100%

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm ^3

Hepatic

* AST and ALT < 2.5 times upper limit of normal (ULN)
* Bilirubin < 1.5 times ULN

Renal

* Creatinine < 1.5 times ULN

Cardiovascular

* Clinically normal cardiac function
* No ischemic heart disease within the past 12 months
* No New York Heart Association grade III or IV cardiac insufficiency
* No unstable angina
* No arryhthmia

Pulmonary

* DLCO > 70% of predicted (for patients randomized to receive erlotinib [arm I] or carmustine [arm II])
* No history of pulmonary disease that would affect pulmonary function including any of the following:

  * Chronic bronchopneumopathy
  * Pleural effusion
  * Interstitial pnuemonia
  * Pulmonary lymphangitis

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after study participation
* No other malignancy except cone biopsied carcinoma of the cervix or adequately treated basal cell or squamous cell skin cancer
* No psychological, familial, sociological, or geographical factors that would preclude study compliance

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior HER-targeted agents
* No concurrent growth factors for neutrophil count elevation
* No concurrent epoetin alfa

Chemotherapy

* Prior adjuvant temozolomide allowed
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas)
* No more than 1 prior adjuvant chemotherapy regimen
* No prior chemotherapy for recurrent disease

Endocrine therapy

* Must be on a stable or decreasing dose of corticosteroids for at least 2 weeks before study entry

Radiotherapy

* See Disease Characteristics
* More than 3 months since prior radiotherapy to the brain
* No prior high-dose radiotherapy (> 65 Gy), stereotactic radiosurgery, or internal radiotherapy unless disease recurrence confirmed

Surgery

* See Disease Characteristics

Other

* No prior participation in experimental therapies
* No concurrent CYP3A4 inhibitors (e.g., ketoconazole, erythromycin, troleandomycin, cimetidine, or grapefruit juice)
* No concurrent warfarin or other coumarin derivatives

  * Concurrent low-molecular weight heparin allowed
* No other concurrent investigational drugs

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2004-05; Primary Completion 2006-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Progression-free survival at 6 months

SECONDARY OUTCOMES:
Response (complete [CR] or partial response [PR]) measured by McDonald's criteria at least 4 weeks after first documented response and every 8 weeks until disease progression or until start of another treatment
Severe toxic events assessed by CTCAE v3.0 at the end of each course
Progression-free survival at 1 year
Overall survival at 6 months and 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Martin J. van Den Bent, MD, Study Chair — Daniel Den Hoed Cancer Center at Erasmus Medical Center
Locations (10):
- U.Z. Gasthuisberg, Leuven, Belgium
- France (5):
  - Centre de Lutte Contre le Cancer Georges-Francois Leclerc, Dijon
  - Centre Regional Rene Gauducheau, Nantes-Saint Herblain
  - Centre Antoine Lacassagne, Nice
  - CHU Pitie-Salpetriere, Paris
  - Institut Gustave Roussy, Villejuif
- Azienda Ospedaliera di Padova, Padua, Italy
- Netherlands (2):
  - University Medical Center Rotterdam at Erasmus Medical Center, Rotterdam
  - Medisch Centrum Haaglanden, The Hague
- Western Infirmary, Glasgow, Scotland, United Kingdom

REFERENCES:
- [Result] van den Bent MJ, Brandes AA, Rampling R, Kouwenhoven MC, Kros JM, Carpentier AF, Clement PM, Frenay M, Campone M, Baurain JF, Armand JP, Taphoorn MJ, Tosoni A, Kletzl H, Klughammer B, Lacombe D, Gorlia T. Randomized phase II trial of erlotinib versus temozolomide or carmustine in recurrent glioblastoma: EORTC brain tumor group study 26034. J Clin Oncol. 2009 Mar 10;27(8):1268-74. doi: 10.1200/JCO.2008.17.5984. Epub 2009 Feb 9. PMID 19204207
- [Result] van den Bent MJ, Brandes A, Rampling R, et al.: Randomized phase II trial of erlotinib (E) versus temozolomide (TMZ) or BCNU in recurrent glioblastoma multiforme (GBM): EORTC 26034. [Abstract] J Clin Oncol 25 (Suppl 18): A-2005, 2007.